CLINICAL TRIAL: NCT01854918
Title: A Multicenter, Controlled, Open-label Extension (OLE) Study to Assess the Long-term Safety and Efficacy of AMG 145
Brief Title: Open-label Extension Study of Evolocumab (AMG 145) in Adults With Hyperlipidemia and Mixed Dyslipidemia
Acronym: OSLER-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120138; 2012-004357-83 (EudraCT Number)
Record Dates: First submitted 2013-05-01; First posted 2013-05-16 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Hyperlipidemia and Mixed Dyslipidemia
Keywords: High cholesterol; Raised cholesterol; Cholesterol; Elevated Cholesterol
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia | interventions — evolocumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (Active Comparator): Participants received standard of care (SOC) treatment for the first year of the study (SOC-controlled period). At week 48, participants began treatment with evolocumab at a dose of either 140 mg every 2 weeks (Q2W) or 420 mg every month (QM), based on participant choice, for approximately 2 years during the all-investigational product [all-IP] period.
  Interventions: Biological: Evolocumab; Drug: Standard of Care
- Evolocumab + Standard of Care (Experimental): Participants received subcutaneous evolocumab plus standard of care during the first year of the study (SOC-controlled period) and for approximately 2 years during the all-IP period. Evolocumab was administered at a dose of 140 mg every 2 weeks (Q2W) or 420 mg every month (QM) based on participant choice.
  Interventions: Biological: Evolocumab; Drug: Standard of Care

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection either every 2 weeks or once a month (patient preference) using a prefilled autoinjector pen
  Other Names: AMG 145; Repatha
Drug: Standard of Care — Standard of care therapy as per local practices. This could include prescribed therapies and/or dietary/exercise regimes

SUMMARY:
This study will contribute to the evaluation of long-term safety, tolerability and efficacy of evolocumab (AMG 145) in adults with hyperlipidemia and adults with mixed dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

- Complete a qualifying evolocumab (AMG 145) parent study (ie, Study 20110114 [NCT01763827], 20110115 [NCT01763866], 20110116 [NCT01763905], 20110117 [NCT01763918], 20110109 [NCT01516879], 20120122 [NCT01953328], 20120332 [NCT01984424], 20120348 [NCT01849497], or 20120356 [NCT01879319]).

Exclusion Criteria:

* Experienced a treatment-related serious adverse event that led to study drug discontinuation in the parent study
* Have an unstable medical condition, in the judgment of the investigator
* Known sensitivity to any of the products to be administered during dosing
* Currently enrolled in another investigational device or drug study (excluding evolocumab (AMG 145) parent study), or less than 30 days since ending another investigational device or drug study(s),or receiving other investigational agent(s)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3681 (Actual)
Dates: Start 2013-04-23 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (310):
- United States (97):
  - Research Site, Birmingham, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Beverly Hills, California
  - Research Site, Carmichael, California
  - Research Site, Encinitas, California
  - Research Site, Huntington Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Newport Beach, California
  - Research Site, San Diego, California
  - Research Site, Santa Ana, California
  - Research Site, Santa Rosa, California
  - Research Site, Spring Valley, California
  - Research Site, Thousand Oaks, California
  - Research Site, Torrance, California
  - Research Site, Tustin, California
  - Research Site, Ventura, California
  - Research Site, Littleton, Colorado
  - Research Site, Daytona Beach, Florida
  - Research Site, DeLand, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Ponte Vedra, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Sanford, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Sterling, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Monroe, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Portland, Maine
  - Research Site, Bethesda, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Ayer, Massachusetts
  - Research Site, Quincy, Massachusetts
  - Research Site, Ypsilanti, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, Olive Branch, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Endwell, New York
  - Research Site, Manlius, New York
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Williamsville, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Cadiz, Ohio
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Mansfield, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Sandusky, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Hillsboro, Oregon
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Lansdale, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Jackson, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Suffolk, Virginia
  - Research Site, Renton, Washington
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
- Australia (12):
  - Research Site, Camperdown, New South Wales
  - Research Site, Maroubra, New South Wales
  - Research Site, Sydney, New South Wales
  - Research Site, Auchenflower, Queensland
  - Research Site, Carina Heights, Queensland
  - Research Site, Sherwood, Queensland
  - Research Site, Woolloongabba, Queensland
  - Research Site, Ashford, South Australia
  - Research Site, Fullarton, South Australia
  - Research Site, Heidelberg Heights, Victoria
  - Research Site, Melbourne, Victoria
  - Research Site, Perth, Western Australia
- Research Site, Salzburg, Austria
- Belgium (16):
  - Research Site, Anthée
  - Research Site, Blankenberge
  - Research Site, Brussels
  - Research Site, Chênée
  - Research Site, Ghent
  - Research Site, Gozée
  - Research Site, Gribomont
  - Research Site, Halen
  - Research Site, Ham
  - Research Site, Hasselt
  - Research Site, La Louvière
  - Research Site, Linkebeek
  - Research Site, Ostend
  - Research Site, Tessenderlo
  - Research Site, Tremelo
  - Research Site, Vilvoorde
- Canada (23):
  - Research Site, Burnaby, British Columbia
  - Research Site, Kelowna, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Cambridge, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Woodstock, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Granby, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Lachine, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
- Czechia (12):
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, Hradec Králové
  - Research Site, Kladno
  - Research Site, Litoměřice
  - Research Site, Moravské Budějovice
  - Research Site, Olomouc
  - Research Site, Pardubice
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Slaný
  - Research Site, Svitavy
- Denmark (5):
  - Research Site, Aalborg
  - Research Site, Aarhus N
  - Research Site, Ballerup Municipality
  - Research Site, Glostrup Municipality
  - Research Site, Vejle
- France (8):
  - Research Site, Brest
  - Research Site, Bron
  - Research Site, Caen
  - Research Site, Dijon
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Vénissieux
- Germany (12):
  - Research Site, Bad Krozingen
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Hellersdorf
  - Research Site, Heppenheim an der Bergstrasse
  - Research Site, Homburg
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, Messkirch
  - Research Site, München
  - Research Site, Witten
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, New Territories
- Hungary (11):
  - Research Site, Baja
  - Research Site, Berettyóújfalu
  - Research Site, Budapest
  - Research Site, Eger
  - Research Site, Gyöngyös
  - Research Site, Hódmezővásárhely
  - Research Site, Jászberény
  - Research Site, Komárom
  - Research Site, Mosonmagyaróvár
  - Research Site, Pécs
  - Research Site, Szeged
- Italy (11):
  - Research Site, Bologna
  - Research Site, Cagliari
  - Research Site, Chieti
  - Research Site, Cinisello Balsamo (MI)
  - Research Site, Ferrara
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Trieste
- Japan (31):
  - Research Site, Noda, Chiba
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kitakyusyu-shi, Fukuoka
  - Research Site, Koriyama-shi, Fukushima
  - Research Site, Maebashi, Gunma
  - Research Site, Takasaki-shi, Gunma
  - Research Site, Sapporo, Hokkaido
  - Research Site, Tsuchiura-shi, Ibaraki
  - Research Site, Morioka, Iwate
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Tomigusuku-shi, Okinawa
  - Research Site, Ibaraki-shi, Osaka
  - Research Site, Toyonaka-shi, Osaka
  - Research Site, Koshigaya-shi, Saitama
  - Research Site, Niiza-shi, Saitama
  - Research Site, Arakawa-ku, Tokyo
  - Research Site, Chiyoda-ku, Tokyo
  - Research Site, Chofu-shi, Tokyo
  - Research Site, Edogawa-ku, Tokyo
  - Research Site, Hachioji-shi, Tokyo
  - Research Site, Katsushika-ku, Tokyo
  - Research Site, Koto-ku, Tokyo
  - Research Site, Minato-ku, Tokyo
  - Research Site, Ōta-ku, Tokyo
  - Research Site, Setagaya-ku, Tokyo
  - Research Site, Shibuya-ku, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Toshima-ku, Tokyo
- Netherlands (11):
  - Research Site, Amsterdam
  - Research Site, Den Helder
  - Research Site, Groningen
  - Research Site, Hoogeveen
  - Research Site, Hoorn
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Tilburg
  - Research Site, Utrecht
  - Research Site, Waalwijk
  - Research Site, Zwijndrecht
- Research Site, Christchurch, New Zealand
- Norway (2):
  - Research Site, Ålesund
  - Research Site, Oslo
- Research Site, Lodz, Poland
- Russia (6):
  - Research Site, Barnaul
  - Research Site, Kemerovo
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Saratov
- South Africa (10):
  - Research Site, Centurion, Gauteng
  - Research Site, Johannesburg, Gauteng
  - Research Site, Midrand, Gauteng
  - Research Site, Sunninghill, Gauteng
  - Research Site, eManzimtoti, KwaZulu-Natal
  - Research Site, Observatory, Western Cape
  - Research Site, Paarl, Western Cape
  - Research Site, Parow, Western Cape
  - Research Site, Somerset West, Western Cape
  - Research Site, Bloemfontein
- Research Site, Seoul, South Korea
- Spain (5):
  - Research Site, Córdoba, Andalusia
  - Research Site, Zaragoza, Aragon
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, Reus, Catalonia
  - Research Site, Madrid
- Sweden (5):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Örebro
  - Research Site, Stockholm
  - Research Site, Uddevalla
- Switzerland (8):
  - Research Site, Bellinzona
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Lugano
  - Research Site, Muensterlingen
  - Research Site, Reinach
  - Research Site, Sankt Gallen
  - Research Site, Zurich
- Taiwan (2):
  - Research Site, Kaohsiung City
  - Research Site, Taipei
- United Kingdom (17):
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, Cardiff
  - Research Site, Chesterfield
  - Research Site, Chorley
  - Research Site, Coventry
  - Research Site, Doncaster
  - Research Site, Glasgow
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Reading
  - Research Site, Telford
  - Research Site, Wakefield
  - Research Site, West Bromwich
  - Research Site, Whitby

REFERENCES:
- [Background] Kasichayanula S, Grover A, Emery MG, Gibbs MA, Somaratne R, Wasserman SM, Gibbs JP. Clinical Pharmacokinetics and Pharmacodynamics of Evolocumab, a PCSK9 Inhibitor. Clin Pharmacokinet. 2018 Jul;57(7):769-779. doi: 10.1007/s40262-017-0620-7. PMID 29353350
- [Result] Sattar N, Toth PP, Blom DJ, Koren MJ, Soran H, Uhart M, Elliott M, Cyrille M, Somaratne R, Preiss D. Effect of the Proprotein Convertase Subtilisin/Kexin Type 9 Inhibitor Evolocumab on Glycemia, Body Weight, and New-Onset Diabetes Mellitus. Am J Cardiol. 2017 Nov 1;120(9):1521-1527. doi: 10.1016/j.amjcard.2017.07.047. Epub 2017 Jul 31. PMID 28844508
- [Result] Hovingh GK, Raal FJ, Dent R, Stefanutti C, Descamps O, Masana L, Lira A, Bridges I, Coll B, Sullivan D. Long-term safety, tolerability, and efficacy of evolocumab in patients with heterozygous familial hypercholesterolemia. J Clin Lipidol. 2017 Nov-Dec;11(6):1448-1457. doi: 10.1016/j.jacl.2017.09.003. Epub 2017 Sep 22. PMID 29066265
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867
- [Derived] Sabatine MS, Giugliano RP, Wiviott SD, Raal FJ, Blom DJ, Robinson J, Ballantyne CM, Somaratne R, Legg J, Wasserman SM, Scott R, Koren MJ, Stein EA; Open-Label Study of Long-Term Evaluation against LDL Cholesterol (OSLER) Investigators. Efficacy and safety of evolocumab in reducing lipids and cardiovascular events. N Engl J Med. 2015 Apr 16;372(16):1500-9. doi: 10.1056/NEJMoa1500858. Epub 2015 Mar 15. PMID 25773607
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 365 study centers in 24 countries in Europe, North America, and Asia Pacific from 23 April 2013 to 31 August 2015.
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive evolocumab plus standard of care (SOC) or SOC alone for the first year. In years 2 and 3 all participants received evolocumab. Randomization was stratified by the parent study and parent study dose frequency (every 2 weeks [Q2W] or once monthly [QM]).
Period: SOC-controlled Period (Year 1)
Arm/Group | Standard of Care | Evolocumab + Standard of Care
Started | 1227 | 2454
Received Evolocumab | 5 (5 participants received evolocumab in error) | 2452
Completed | 1197 | 2391
Not Completed | 30 | 63
Not completed — Withdrawal by Subject | 20 | 49
Not completed — Decision by Sponsor | 2 | 1
Not completed — Lost to Follow-up | 3 | 8
Not completed — Death | 5 | 5
Period: All-IP Period (Years 2 and 3)
Arm/Group | Standard of Care | Evolocumab + Standard of Care
Started | 1197 | 2391
Received Evolocumab | 1152 | 2291
Completed | 1079 | 2196
Not Completed | 118 | 195
Not completed — Withdrawal by Subject | 78 | 117
Not completed — Decision by Sponsor | 8 | 11
Not completed — Lost to Follow-up | 27 | 51
Not completed — Death | 5 | 16

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Evolocumab + Standard of Care | Total
Number analyzed (Participants) | 1227 | 2454 | 3681
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (10.7) | 58.6 (10.7) | 58.7 (10.7)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 823 | 1665 | 2488
  ≥ 65 years | 404 | 789 | 1193
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 560 | 1176 | 1736
  Male | 667 | 1278 | 1945
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58 | 109 | 167
  Not Hispanic or Latino | 1169 | 2345 | 3514
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 5 | 7
  Asian | 152 | 288 | 440
  Black or African American | 49 | 84 | 133
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  White | 1003 | 2041 | 3044
  Other | 16 | 30 | 46
  Mixed Race | 3 | 4 | 7
Region [Count of Participants; unit: Participants]
  North America | 514 | 1001 | 1515
  Europe | 504 | 1018 | 1522
  Asia Pacific | 209 | 435 | 644
Parent Study Baseline Low-density Lipoprotein Cholesterol (LDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 125.8 (49.3) | 127.4 (51.7) | 126.9 (50.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse event (AE) severity assessments were made using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) grading, version 4.0, where grade 1 = mild AE, grade 2 = moderate AE, Grade 3 = severe AE, grade 4 = life-threatening AE and Grade 5 = death due to AE.
Time Frame: 48 weeks in the SOC-controlled period and up to 2 years in the All-IP period
Population: All randomized participants (year 1) and randomized participants on study and who received at least 1 dose of evolocumab in the all-IP period (years 2-3).
Measure: Count of Participants; unit: Participants
Groups:
- Year 1: Standard of Care: Participants received standard of care (SOC) treatment for the first year of the study (SOC-controlled period).
- Year 1: Evolocumab + Standard of Care: Participants received subcutaneous evolocumab plus standard of care during the first year of the study (SOC-controlled period). Evolocumab was administered at a dose of 140 mg every 2 weeks (Q2W) or 420 mg every month (QM) based on participant choice.
- Years 2-3: SOC / Evolocumab + SOC: At week 48, participants began treatment with evolocumab at a dose of either 140 mg Q2W or 420 mg QM, based on participant choice, plus SOC, for approximately 2 years during the all-IP period.
- Years 2-3: Evolocumab + SOC / Evolocumab + SOC: Participants continued to receive evolocumab plus SOC for approximately 2 years during the all-IP period. Evolocumab was administered at a dose of 140 mg Q2W or 420 mg QM based on participant choice.
Arm/Group | Year 1: Standard of Care | Year 1: Evolocumab + Standard of Care | Years 2-3: SOC / Evolocumab + SOC | Years 2-3: Evolocumab + SOC / Evolocumab + SOC
Number analyzed (Participants) | 1227 | 2454 | 1152 | 2291
Participants
  All adverse events | 796 | 1655 | 929 | 1789
  Adverse events ≥ grade 2 | 519 | 1070 | 700 | 1339
  Adverse events ≥ grade 3 | 124 | 225 | 214 | 379
  Adverse events ≥ grade 4 | 7 | 17 | 11 | 35
  Serious adverse events | 104 | 195 | 178 | 332
  AEs leading to discontinuation of evolocumab | 0 | 55 | 26 | 42
  Fatal adverse events | 5 | 5 | 3 | 16
  Device related adverse events | 0 | 57 | 25 | 45

2. Secondary Outcome: Percent Change From Baseline in LDL-C at Weeks 48 and 104
Time Frame: Baseline of the parent study and weeks 48 amd 104
Population: Participants who were randomized in 20120138 and on-study and with known dosing information in the All-IP period, and with non-missing data at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Standard of Care | Evolocumab + Standard of Care
Number analyzed (Participants) | 1152 | 2291
percent change
  Week 48: number analyzed (Participants) | 1115 | 2241
  Week 48 | 7.43 (38.93) | -51.59 (28.88)
  Week 104: number analyzed (Participants) | 1087 | 2166
  Week 104 | -49.96 (33.29) | -50.31 (30.34)

3. Secondary Outcome: Change From Baseline in LDL-C at Weeks 48 and 104
Time Frame: Baseline of the parent study and weeks 48 amd 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Standard of Care | Evolocumab + Standard of Care
Number analyzed (Participants) | 1152 | 2291
mg/dL
  Week 48: number analyzed (Participants) | 1115 | 2241
  Week 48 | 0.4 (43.9) | -68.8 (46.6)
  Week 104: number analyzed (Participants) | 1087 | 2166
  Week 104 | -66.4 (50.1) | -67.2 (46.6)

ADVERSE EVENTS:
Time Frame: 48 weeks in the SOC-controlled period and up to 2 years in the All-IP period.
Description: Adverse evens are reported for all randomized participants in the SOC-controlled period (year 1) and for all participants who entered the all-IP period (years 2-3).
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Years 2-3: Total: All participants in the All-IP period who received evolocumab plus SOC for approximately 2 years. Evolocumab was administered at a dose of 140 mg Q2W or 420 mg QM based on participant choice.
Arm/Group | Year 1: Standard of Care | Year 1: Evolocumab + Standard of Care | Years 2-3: SOC / Evolocumab + SOC | Years 2-3: Evolocumab + SOC / Evolocumab + SOC | Years 2-3: Total
All-Cause Mortality (participants affected / at risk) | 5/1227 | 5/2454 | 5/1197 | 16/2391 | 21/3588
Serious Adverse Events (participants affected / at risk) | 104/1227 | 195/2454 | 181/1197 | 344/2391 | 525/3588
Other Adverse Events (participants affected / at risk) | 334/1227 | 681/2454 | 498/1197 | 928/2391 | 1426/3588
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Year 1: Standard of Care (N=1227) | Year 1: Evolocumab + Standard of Care (N=2454) | Years 2-3: SOC / Evolocumab + SOC (N=1197) | Years 2-3: Evolocumab + SOC / Evolocumab + SOC (N=2391) | Years 2-3: Total (N=3588)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 2
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 4 | 8 | 3 | 12 | 15
Angina pectoris (Cardiac disorders) | 0 | 7 | 10 | 8 | 18
Angina unstable (Cardiac disorders) | 6 | 7 | 4 | 11 | 15
Aortic valve disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Aortic valve sclerosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1 | 7 | 7 | 14
Atrial flutter (Cardiac disorders) | 1 | 1 | 0 | 3 | 3
Atrioventricular block (Cardiac disorders) | 1 | 0 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 2
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 4 | 4
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | 2 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 3 | 6 | 9
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 4 | 3 | 2 | 7 | 9
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 2 | 1 | 3 | 4
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 5 | 0 | 2 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 4 | 5
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1 | 2
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Rheumatic heart disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 2 | 1 | 3
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 2 | 0 | 2 | 2
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0 | 1
Hyperparathyroidism primary (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Blindness transient (Eye disorders) | 0 | 0 | 1 | 0 | 1
Cataract (Eye disorders) | 1 | 1 | 1 | 0 | 1
Macular fibrosis (Eye disorders) | 0 | 0 | 1 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Anal skin tags (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 3
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 4
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 4
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 3
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 2 | 3 | 3 | 6
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Large intestine polyp (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 4
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Short-bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 1 | 3 | 4 | 7
Complication associated with device (General disorders) | 0 | 0 | 0 | 1 | 1
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 2 | 1 | 1 | 2
Impaired healing (General disorders) | 0 | 0 | 1 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 1 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 4 | 10 | 8 | 18
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Polyp (General disorders) | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 2
Sudden death (General disorders) | 1 | 1 | 0 | 0 | 0
Vascular stent occlusion (General disorders) | 0 | 0 | 0 | 1 | 1
Vascular stent stenosis (General disorders) | 1 | 1 | 0 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 3 | 3 | 6
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 3 | 3 | 6
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 3 | 5 | 0 | 5
Gallbladder necrosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0
Non-alcoholic fatty liver (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Allergy to arthropod sting (Immune system disorders) | 0 | 2 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 1 | 1
Contrast media allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Abscess jaw (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Abscess neck (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 1 | 3 | 4
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 2 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 3 | 3 | 6
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 2 | 1 | 2 | 5 | 7
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Epididymitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Hepatitis B (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 2 | 3
Intervertebral discitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Neurosyphilis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 4 | 12 | 16
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Postoperative abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 1 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1 | 1 | 2
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 2
Urosepsis (Infections and infestations) | 0 | 2 | 0 | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Anastomotic complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 2 | 4
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 2
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 3
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 2 | 3
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4 | 4
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 2
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
VIIIth nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Vascular graft stenosis (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Anticoagulation drug level below therapeutic (Investigations) | 0 | 0 | 1 | 0 | 1
Antimitochondrial antibody positive (Investigations) | 0 | 0 | 1 | 0 | 1
Antinuclear antibody (Investigations) | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood immunoglobulin M increased (Investigations) | 0 | 0 | 1 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 1 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 1
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 1 | 0 | 1
Scan myocardial perfusion abnormal (Investigations) | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5 | 5
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 2 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Diffuse idiopathic skeletal hyperostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 3
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 6 | 6 | 12
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 4 | 6
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 12 | 22 | 22 | 44
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 4
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 4 | 5
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 1 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 2
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1 | 2
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2 | 4
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1 | 2
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 2
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Papillary tumour of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Penile neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 3 | 4 | 7
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3 | 3
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Testicular seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Ataxia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 2 | 0 | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 1 | 7 | 8
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 2
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemic seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 1 | 0 | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Myelopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Nerve root compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Paresis (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 4 | 4
Sciatica (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0 | 2 | 2
Spinal cord haematoma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 3 | 1 | 2 | 5 | 7
Transient global amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 3 | 0 | 3 | 5 | 8
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Visual field defect (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Device leakage (Product Issues) | 0 | 0 | 0 | 1 | 1
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Agoraphobia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1
Bipolar I disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 1 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 4 | 4
Drug dependence (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 3
Bladder fibrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 1 | 2 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 4 | 1 | 4 | 5
Renal artery stenosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Renal infarct (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 2
Ureteral spasm (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 3 | 0 | 2 | 2
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 2 | 3 | 2 | 5
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
Genital prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Mastoptosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 2
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 1
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 1
Rectocele (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 1
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3 | 5
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 4 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 4 | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 2 | 1 | 1 | 2
Aortic dilatation (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 4 | 0 | 4
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Artery dissection (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 1 | 1
Hypertension (Vascular disorders) | 2 | 1 | 1 | 4 | 5
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 1 | 1
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Labile blood pressure (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Malignant hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Microangiopathy (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 2 | 0 | 2
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 2 | 0 | 1 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 1 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Subclavian artery stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 2 | 2
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Year 1: Standard of Care (N=1227) | Year 1: Evolocumab + Standard of Care (N=2454) | Years 2-3: SOC / Evolocumab + SOC (N=1197) | Years 2-3: Evolocumab + SOC / Evolocumab + SOC (N=2391) | Years 2-3: Total (N=3588)
Bronchitis (Infections and infestations) | 43 | 78 | 70 | 132 | 202
Influenza (Infections and infestations) | 28 | 66 | 60 | 115 | 175
Nasopharyngitis (Infections and infestations) | 108 | 201 | 151 | 253 | 404
Upper respiratory tract infection (Infections and infestations) | 55 | 104 | 99 | 178 | 277
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 | 106 | 80 | 162 | 242
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 83 | 78 | 147 | 225
Myalgia (Musculoskeletal and connective tissue disorders) | 43 | 88 | 61 | 67 | 128
Hypertension (Vascular disorders) | 56 | 87 | 78 | 180 | 258

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2015-04-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT01854918/Prot_000.pdf
  • Statistical Analysis Plan (2013-11-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT01854918/SAP_001.pdf